CLINICAL TRIAL: NCT05083611
Title: The Effectiveness of Graded Motor Imagery in Phantom Limb Pain in Amputee Patients (GraMI Protocol)
Brief Title: Graded Motor Imagery in Phantom Limb Pain (GraMI Protocol)
Acronym: GraMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Principal Investigator, Sandra Rierola Fochs, Physiotherapist, University of Vic - Central University of Catalonia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTGraMI01
Record Dates: First submitted 2021-10-01; First posted 2021-10-19 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Phantom Limb Pain
Keywords: Phantom limb pain; Graded motor imagery; Treatment; Amputee
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive an information session on phantom limb pain (1 hour) and will continue with the usual treatment received.
- Experimental group (Experimental): The experimental group will receive an educational session on phantom limb pain and the previously designed GraMI protocol through a systematic review and validation through a study with Delphi methodology. This protocol contains the three techniques with their defined intensity, frequency, duration and progression.
  Interventions: Other: GraMI

INTERVENTIONS:
Other: GraMI — The intervention will last 6 weeks. Each technique lasts for 2 weeks. The first two techniques will be performed through the previously designed mobile application and the last technique will be performed through a mirror box. The patient can do it autonomously with the supervision of the principal investigator.
  Arms: Experimental group

SUMMARY:
The International Association for the Study of Pain defines phantom limb pain (PLP) as that pain referred to a part of the body that has been previously removed as if it were still present. It affects between 55-80% of the population who has suffered an amputation, but not in the same frequency and intensity. Graded motor imagery (GMI) is a progressive, physiotherapeutic treatment modality developed to train and reorganize the brain based on three consecutive techniques: laterality recognition, motor imagery, and mirror therapy. The scientific evidence on the implementation of GMI in PLP is scarce, noting that there is no standardized way to use it in this patient profile. Therefore, the need is generated to develop and validate a GMI protocol to address the PLP and test its effectiveness.

The study hypothesis is that graded motor imagery is a conservative treatment method based on motor learning, neuroplasticity, and mirror neuron stimulation that may have positive effects in decreasing phantom limb pain in the amputated patient, and as a consequence, decrease the associated psychological factors and improve the quality of life and functionality of the person.

A randomized clinical trial will be performed with simple blinding, following the CONSORT guide for this type of study.

It will be carried out at the community level with supervision and follow-up by the principal investigator.

DETAILED DESCRIPTION:
The International Association for the Study of Pain defines phantom limb pain (PLP) as that pain referred to a part of the body that has been previously removed as if it were still present. It affects between 55-80% of the population who has suffered an amputation, but not in the same frequency and intensity. The persistence of this pain over time may decrease the person's quality of life. The main hypothesis is that after an amputation, maladaptive plasticity occurs at the level of the primary motor and sensory cortex, causing an incongruity of visual, motor and sensory information.

Graded motor imagery (GMI) is a progressive, physiotherapeutic treatment modality developed to train and reorganize the brain based on three consecutive techniques: laterality recognition, motor imagery, and mirror therapy. The scientific evidence on the implementation of GMI in PLP is scarce, noting that there is no standardized way to use it in this patient profile. Therefore, the need is generated to develop and validate a GMI protocol to address the PLP and test its effectiveness.

Therefore, at the beginning of this project, a systematic review was performed to know the effectiveness of the GMI, and the techniques that make it up, on the PLP of the amputated patient, and thus be able to design an GMI protocol based on scientific evidence. Subsequently, this protocol was validated through a group of international experts through a study with Delphi methodology, resulting in the GMI protocol called GraMI.

The GraMI protocol is easy to implement, allowing the patient to perform it autonomously at home with the follow-up of a professional. It is necessary to have a mirror box and a mobile application to be able to carry out the intervention. During the COVID-19 pandemic, many patients remained in their homes confined without being able to access their rehabilitation, which caused alterations in the quality of life, in the prescribed treatment and in the evolution of the symptoms. The promotion of the patient's self-care at home, enhances their active participation and the intensity of the intervention, so that greater benefits can be obtained and consequently improvement in the quality of life.

Objectives:

Main objective:

- Study the effects of the GraMI protocol on DMF in the amputee patient.

Secondary objectives:

* Design a mobile application to be able to carry out the intervention and determine its usability.
* Analyse the effects of the GraMI protocol on the quality of life, functionality and psychological aspects of amputee patients.
* Understand the perception and satisfaction obtained through the intervention.

A randomized clinical trial will be performed with simple blinding, following the CONSORT guide for this type of study.

It will be carried out at the community level with supervision and follow-up by the principal investigator.

During recruitment, a person outside the intervention will randomize the participants through sealed envelopes where they will be assigned to the control group or intervention group. A non-probabilistic sampling type for quotas will be used.

The intervention of the two groups will last 9 weeks plus 12 weeks of follow-up. During the study, three assessments will be performed, one at the beginning, one after the intervention (9 weeks) and one follow-up (12 weeks post-intervention).

These assessments will collect quantitative variables and also conduct semi-structured individual interviews with participants who are part of the intervention group in order to know and understand the influence of phantom limb pain in their lives and the degree of satisfaction obtained through the intervention.

ELIGIBILITY:
Inclusion Criteria:

* People over the age 18.
* Amputation of a limb.
* Minimum score of 3 on the VAS.
* Under pharmacological treatment for pain
* Pharmacologically stable.
* Be discharged from hospital.

Exclusion Criteria:

* Visual disturbances (hemianopia).
* Significant neurological or cognitive disturbances (attention deficit, sensory aphasia).
* Receive two of the three techniques that make up the GMI as treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline phantom limb pain at 9 weeks post-intervention and 12 weeks follow-up | Post intervention (9 weeks) and 12 weeks follow-up
  Assessed by Short Form McGill Pain Questionnaire. Assesses pain qualitatively and quantitatively, it is a self-testifying scale. It consists of 15 pain descriptors, of which 11 are sensitive categories and 4 affective. In addition, it contains an analog visual scale of pain. It is self-contesting and each descriptor has three columns (medium, moderate, severe), where the patient must mark the degree to which that descriptor persists in their pain, in case of not being present they can leave it blank. . Columns are categorized to be 0; no pain, 1; mig, 2; moderate, 3; severe. The higher the score the more pain it indicates

SECONDARY OUTCOMES:
Change from quality of life at 9 weeks post-intervention and 12 weeks follow-up | Post intervention (9 weeks) and 12 weeks follow-up
  Assessed by EuroQol scale. It is a self-challenging scale made up of 5 dimensions: mobility, self-care, regular activities, pain / discomfort and anxiety / depression. Each dimension has 5 levels: no problems, mild, moderate, severe and extreme problems. The patient is asked to indicate his / her state of health by ticking the box together with the most appropriate statement in each of the 5 dimensions. In addition, it contains a numerical scale from 0 to 100 to quantify the degree of health status on the day of assessment.
Change from baseline functionality at 9 weeks post-intervention and 12 weeks follow-up | Post intervention (9 weeks) and 12 weeks follow-up
  Assessed by Functional Independence Scale (FIM). It is a scale built from 18 items within 6 areas of operation: personal care, sphincter control, mobility, walking, communication and social knowledge.
  The maximum score for each item is 7 and the minimum is 1.
Change from baseline physcological aspects at 9 weeks post-intervention and 12 weeks follow-up | Post intervention (9 weeks) and 12 weeks follow-up
  Assessed by Beck depression inventory. It is a self-answering scale of 21 questions. Each question is graded on a 4-point scale ranging from 0 to 3, with 0 experiencing no symptoms and 3 experiencing symptoms severely.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Rierola Fochs, Principal Investigator — Universitat de Vic- Universitat Central de Catalunya (UVic-UCC)
Locations (1):
- Sandra Rierola Fochs, Vic, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Anaforoglu Kulunkoglu B, Erbahceci F, Alkan A. A comparison of the effects of mirror therapy and phantom exercises on phantom limb pain. Turk J Med Sci. 2019 Feb 11;49(1):101-109. doi: 10.3906/sag-1712-166. PMID 30762318
- [Background] Limakatso K, Corten L, Parker R. The effects of graded motor imagery and its components on phantom limb pain and disability in upper and lower limb amputees: a systematic review protocol. Syst Rev. 2016 Sep 1;5(1):145. doi: 10.1186/s13643-016-0322-5. PMID 27582042
- [Background] Moseley GL. Graded motor imagery for pathologic pain: a randomized controlled trial. Neurology. 2006 Dec 26;67(12):2129-34. doi: 10.1212/01.wnl.0000249112.56935.32. Epub 2006 Nov 2. PMID 17082465
- [Background] Limakatso K, Madden VJ, Manie S, Parker R. The effectiveness of graded motor imagery for reducing phantom limb pain in amputees: a randomised controlled trial. Physiotherapy. 2020 Dec;109:65-74. doi: 10.1016/j.physio.2019.06.009. Epub 2019 Jun 28. PMID 31992445
- [Derived] Rierola-Fochs S, Terradas-Monllor M, Grau-Carrion S, Ochandorena-Acha M, Minobes-Molina E, Merchan-Baeza JA. Graded Motor Imagery (GRAMI Protocol) for Phantom Limb Pain: A Randomised Clinical Trial of Home-Based Intervention. Eur J Pain. 2026 Jan;30(1):e70167. doi: 10.1002/ejp.70167. PMID 41255083
- [Derived] Rierola-Fochs S, Merchan-Baeza JA, Minobes-Molina E. Effectiveness of graded motor imagery protocol in phantom limb pain in amputed patient: Protocol of a randomized clinical trial. PLoS One. 2022 Aug 25;17(8):e0273356. doi: 10.1371/journal.pone.0273356. eCollection 2022. PMID 36006951